CLINICAL TRIAL: NCT07387146
Title: Community Health Worker Navigation to Support Mental Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Riverside (Other)
Collaborators: Cultura y Arte Nativa de las Americas (CANA) (Unknown); Native American Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: OT2OD035895 (NIH)
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Stress; Service Utilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-List Control Arm - Treatment as Usual (No Intervention): Promotora Support for Cultural Healing Practices: Participants assigned to the wait-list control condition will receive standard promotora support as typically provided through CANA's Indigenous Peoples Cultural Arts Healing Center and the Native American Health Center (NAHC), which may include general health promotion, wellness education, and linkage to cultural healing resources. After completing the 12-week wait-list period and follow-up assessment, participants in this group will be offered the full CAPAZ protocolized navigation intervention.
- Protocolized Promotora-Led Navigation (Experimental)
  Interventions: Behavioral: Protocolized Promotora-Led Navigation

INTERVENTIONS:
Behavioral: Protocolized Promotora-Led Navigation — Participants in this group will receive the CAPAZ protocolized navigation intervention, in which trained promotoras-supported by the Lead Study Navigator and the Principal Investigator (PI)-deliver structured, individualized health navigation. The intervention will follow a defined protocol that includes behavioral health screening, care coordination, and facilitated referrals to mental health services, primary care, and social-cultural or community resources as needed. The model also allows participants to integrate cultural and traditional healing practices into their care plan. Each participant will receive up to six promotora sessions over 12 weeks, focusing on improving access to care, stress reduction, and overall wellbeing.
  Arms: Protocolized Promotora-Led Navigation

SUMMARY:
This pilot study tests the feasibility and preliminary impact of a protocolized promotora-led navigation intervention to improve behavioral health access among Latinx and Native American underserved adults. The study is embedded within a community cultural center, leveraging a trusted and culturally grounded environment for recruitment and intervention delivery. Participants will be randomized 1:1 to receive either the promotora navigation intervention or a treatment-as-usual (TAU) condition consisting of cultural resources and promotora-supported wait-list control. The TAU group will continue to receive any usual care during the study period and will be offered the protocolized navigation intervention after completing follow-up assessments. Primary outcomes include feasibility, acceptability, and preliminary changes in behavioral health access, stress reduction, self-efficacy, and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older

  * Speak either English or Spanish
  * Report moderate or higher perceived stress, defined as scoring 14 or above on the Perceived Stress Scale (PSS)

Exclusion Criteria:

* Score below 14 on the Perceived Stress Scale (PSS), indicating low perceived stress and ineligibility for enrollment.

Endorse suicidal ideation on PHQ-9 item 9 (any score > 0) and score at moderate to high risk on the Columbia Suicide Severity Rating Scale (C-SSRS) as assessed by the study psychiatrist/PI.

Report verbal or written suicidal ideation to any study team member. Exhibit any indication of suicidality or threats of harm to others reported or observed by research staff.

Score 16 or higher on the AUDIT, indicating severe alcohol use. Score 6 or higher on the DAST-10, indicating severe drug use. Arrive at screening intoxicated, impairing informed consent capacity or ability to participate.

Present to the screening or interview space with any of the following concerning clinical signs:

* Marked emotional dysregulation such that engagement is not feasible
* Significant physical dishevelment suggesting acute impairment
* Apparent intoxication from alcohol or other substances
* Possible hallucinations or other signs of psychosis
* Any indication that psychological status may compromise safe participation Are unable to complete the screening process due to any of the above concerns (screening will be halted and the participant will be referred for appropriate support).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-09-19 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Baseline, Week 12, Week 24
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.
Depression Patient Health Questionnaire-9 (PHQ-9) | Baseline, Week 12, Week 24
  PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.

SECONDARY OUTCOMES:
Generalized Self-Efficacy Scale (GSES) | Baseline, Week 12, and Week 24
  The General Self-Efficacy Scale measures ones perceived self-efficacy or belief in their ability to cope with different situations and accomplish goals. For each item there is a four choice response scoring from 1-4 and then summed to give a total score with the higher the score the higher the individual's sense of self-efficacy. GSE (10 items): 1-4 scale; sum (10-40); higher = greater self-efficacy.
PROMIS General Self-Efficacy Short Form (4a) | Baseline, Weeks 12, and Week 24
  PROMIS GSE (4 items): 1-5 scale; sum or convert to PROMIS T-score.
Services Use and Benefits | Baseline, Week 12, Week 24
  These researcher-designed measure document services used through navigator referral, degree of difficulty in accessing services, and self-rating of perceived improvement. The measure is available in English and Spanish. Purpose: To understand your experiences using community, cultural, and health services, and the benefits of support from a promotora or community health worker (CHW).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfaro A, Alfaro E, Coto E, Gomez C, Montejo D, Pozo H, Pena R, Rivera C, Cibrian JGR, Rodriguez M, Salazar D, Sierra R, Ulloa J, Uribe V, Flores P, Camarena A. Somos Esenciales, We are Essential: Our Mental Health is Essential. Research for, by and of the Latinx Community in the Mission District during the Pandemic. Acad Pediatr. 2024 Jul;24(5S):95-97. doi: 10.1016/j.acap.2024.01.025. PMID 38991816